CLINICAL TRIAL: NCT01957540
Title: Differential Effect of Ticagrelor Versus Prasugrel Maintenance Dose on Endothelial Function of Peripheral Vessels in Patients With Coronary Artery Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, Dimitrios Alexopoulos, Professor, University of Patras
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PATRASCARDIOLOGY-16
Record Dates: First submitted 2013-09-30; First posted 2013-10-08 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Coronary Artery Disease; Endothelial Function
Keywords: ticagrelor; prasugrel; endothelial function
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ticagrelor; Prasugrel Hydrochloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ticagrelor (Experimental): Ticagrelor 90mg bid for 15 days
  Interventions: Drug: Ticagrelor; Drug: Prasugrel
- Prasugrel (Active Comparator): Prasugrel 10mg od for 15 days
  Interventions: Drug: Ticagrelor; Drug: Prasugrel

INTERVENTIONS:
Drug: Ticagrelor
Drug: Prasugrel

SUMMARY:
Ticagrelor administration, whose molecule resembles to adenosine, led to reduction in overall mortality and thrombotic cardiovascular (CV) events when directly compared to clopidogrel in the PLATO trial, implicating possible pleiotropic actions for the drug. It has been shown that ticagrelor increases adenosine concentration, by interfering with its red blood cells' uptake and by inducing the release of ATP which is then converted to adenosine. Recent studies in healthy volunteers and patients with coronary artery disease (CAD) have shown that ticagrelor increases the coronary blood flow in response to intravenous adenosine administration. Ticagrelor administration, in comparison with other P2Y12 inhibitors, may influence the endothelial function, as assessed by the Peripheral Arterial Tonometry method (EndoPAT 2000 system (Itamar Medical, Caesarea, Israel), which is a method for evaluating endothelial dysfunction and has been found to positively correlate with flow mediated dilatation (FMD).

This is prospective, randomized study with a crossover design, which will be conducted in patients with CAD under prasugrel maintenance dose (MD) 10mg once a day for at least a 3-month period. At Day 0 (day of randomization) eligible patients will be assigned to either:

* Ticagrelor 90mg twice a day for the next 15 days or
* Prasugrel 10mg once a day for the next 15 days At Day 0 (before treatment onset)patients wiil be subjected to a baseline peripheral arterial tonometry measurement. Measurement will be repeated at Day 15 and then treatment crossover will be performed for the next 15 days (without an intervening washout period). At Day 30 patients will be subjected again to peripheral arterial tonometry assessment. Peripheral blood sample will be taken from the patients in Day 0 for genotyping control.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-74 years old
2. Patients with stable CAD who have been submitted(?) to percutaneous intervention for Acute Coronary Syndrome and receiving prasugrel MD 10mg once a day for at least the previous 3 months.
3. Patients giving written Informed Consent.

Exclusion Criteria:

1. Acute Coronary Syndrome
2. Contraindication for administration of prasugrel or ticagrelor

   1. Known hypersensitivity to clopidogrel or ticagrelor
   2. Active bleeding (peptic ulcer, intracranial bleeding)
   3. Severe liver impairment
   4. Any previous history of intracranial bleeding or transient ischemic attack or ischemic cerebrovascular event
   5. Treatment with potent CYP3A4 inhibitors (ketoconazole, clarithromycin, nefazodone, ritonavir, atazanavir)
3. Requirement for oral anticoagulant agents prior to the day 30 visit
4. History of gastrointestinal bleeding, genitourinary bleeding or other site abnormal bleeding within the previous 3 months
5. Increased risk for bradyarrhythmias, according to the investigator's evaluation
6. Severe non-controlled chronic obstructive pulmonary disease
7. Creatinine clearance <30ml/min/1.73mm2
8. HbA1c > 10mg/dl

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Reactive Hyperemia Index (RHI) in the 2 subgroups at the end of 2 periods of treatment | 15 days

SECONDARY OUTCOMES:
Percentage of patients with endothelial dysfunction (RHI<1.67) at the end of 2 periods of treatment | 15 days

CONTACTS AND LOCATIONS:
Locations (1):
- Patras University Hospital, Pátrai, Achaia, Greece

REFERENCES:
- [Derived] Xanthopoulou I, Bei I, Bampouri T, Barampoutis N, Moulias A, Davlouros P, Alexopoulos D. Absence of differential effect of ticagrelor versus prasugrel maintenance dose on endothelial function in patients with stable coronary artery disease. Hellenic J Cardiol. 2018 Nov-Dec;59(6):338-343. doi: 10.1016/j.hjc.2017.12.008. Epub 2017 Dec 29. PMID 29292242